CLINICAL TRIAL: NCT06616701
Title: The Impact of Routine Follow-up Contacts After a Pediatric ED Visit for Youth With Suicide Risk: a Randomized Controlled Trial
Brief Title: The Impact of Routine Follow-up Contacts After a Pediatric ED Visit for Youth With Suicide Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00396477
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Suicidal Ideation
Keywords: Suicidal thoughts; Suicidal behaviors; Suicidal risk
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow up call within 5 days (Experimental): Follow up call within 5 days
  Interventions: Behavioral: Follow up call
- Follow up call within 10 days (No Intervention): Follow up call within 10 days

INTERVENTIONS:
Behavioral: Follow up call — As part of the standard of care, caregivers of youths who present to the hospital with suicidal risk receive a follow up call approximately 5-10 business days after the hospital discharge to assist them with any challenges they may encounter in accessing mental health care, including medication access. The intervention group will receive a call 5 days after discharge. The non-intervention group will receive a call 10 days after discharge.
  Arms: Follow up call within 5 days

SUMMARY:
The goal of this clinical trial is to learn if a social work led follow up program helps caregivers of youths with suicide risk access mental health resources.

Primary aims include:

1. To formalize a mental health follow up protocol that assists youths with engagement of mental health services after a hospital visit.
2. To evaluate and standardize the optimal timing for the follow up phone calls.
3. To assess the proportion of patients with suicide risk who connect with community mental health care within a month after a pediatric emergency department (ED) visit at Johns Hopkins Hospital.
4. To assess the proportion of patients with suicide risk who have repeat ED visits within 3 and 6 months.

The primary outcome of interest is the proportion of youths referred to a community provider who successfully connect to community mental health resources 5 to 10 business days after an ED visit. The secondary outcome will involve repeat ED visits within 3 and 6 months.

DETAILED DESCRIPTION:
The month following an ED discharge is a high-risk period for suicide for patients recovering from a suicide attempt and/or experiencing suicidal ideation, making referrals and follow up critically important. Very few hospital systems, if any, have been able to implement policies and practices that ensure patients at risk for suicide are getting the follow up care they need. Patient navigator interventions have demonstrated success in improving health outcomes across a range of conditions including mental health, and moreover, they have been effective in providing practical support and encouragement to aid patients in accessing community mental health services. Navigators are trained and supervised frontline public health personnel who are hired from the same communities as patients and aid patients in accessing health care and social services. They have shared experiences and nuanced understanding of the communities they serve to help facilitate developing rapport and trust with families, which can help mitigate health care inequities. To the investigator's knowledge, there are no published studies that have evaluated the implementation of patient navigators in the pediatric ED to help caregivers of suicidal youths access community mental health resources after an ED visit.

In the pediatric ED at Johns Hopkins, an ad hoc clinical initiative led by social work (SW) was started in September 2022 with efforts focused on following up with caregivers of patients with mental health emergencies who are discharged from the hospital. SW staff have been calling caregivers a few days after an ED visit or hospitalization to assist with barriers such as challenges in connecting with community mental health resources and accessing prescribed medications.

For this research, this follow up program will be standardized and consistent data collection will be implemented. A randomized controlled trial will be conducted to evaluate the efficacy of this intervention. If the results are promising, evaluation of this program would provide preliminary data for a future study for implementation of a patient navigation program to improve mental health service engagement for youths with suicide risk who are discharged from the pediatric ED.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 8 to 21 years old;
* Who present to the emergency department (ED) and are assessed with suicide risk;
* Who are discharged from the Johns Hopkins Hospital (Pediatric inpatient psychiatric unit, Pediatric Day Hospital, or Pediatric ED) with a mental health referral

Exclusion Criteria:

* Patients who were directly transferred to the inpatient psychiatry unit or the Day Hospital from an outside hospital, bypassing the hospital's ED
* Direct admissions, bypassing the hospital's ED

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 401 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Proportion of youths accessing community mental health resources | From enrollment up to 6 months
  The primary outcome of interest is the proportion of youths referred to a community provider who successfully connect to community mental health resources 5 to 10 business days after an ED visit.

SECONDARY OUTCOMES:
Emergency department revisits | From enrollment up to 6 months
  The secondary outcome will involve repeat ED visits within 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hanae Fujii-Rios, MD MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No